CLINICAL TRIAL: NCT01025141
Title: Study of the Efficacy of Skeletal Anchorage (MINISCREW) Compared to Dental Anchorage During Orthodontic Treatment
Brief Title: Efficacy of Skeletal Anchorage (MINISCREW)
Acronym: Minivis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: DENTOS (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P070610
Record Dates: First submitted 2009-09-29; First posted 2009-12-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Tooth Extraction Status Nos
Keywords: MINISCREW; space extraction closure; anchorage; Orthodontic Treatment; Extraction of 2 Maxillary Premolar; closing of extraction space; patient aged from 12 to 50 years old

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MINISCREW (Experimental): device
  Interventions: Device: Skeletal anchorage (MINISCREW)
- Reference (Active Comparator): dental anchorage
  Interventions: Device: dental anchorage

INTERVENTIONS:
Device: Skeletal anchorage (MINISCREW) — Skeletal anchorage
  Other Names: Skeletal anchorage
  Arms: MINISCREW
Device: dental anchorage — dental anchorage (reference)
  Other Names: dental anchorage (reference)
  Arms: Reference

SUMMARY:
The main objective of the investigators' study is to assess the efficacy of a course of treatment using skeletal anchorage (MINISCREW) as compared with treatment involving dental anchorage (reference) during dentofacial orthopedic treatment.

DETAILED DESCRIPTION:
Multicenter prospective study on patients aged between 12 and 50 years, requiring orthodontic treatment with premolar extractions and closure of the extraction spaces by distalization of the 6 anterior teeth. In the experimental group (50 patients) distalization will be performed using skeletal anchorage (MINISCREW). In the control group (50 patients), distalization will be by dental anchorage.

The main evaluation criterion will be extraction space closure after 8 months of treatment. Angle class I cuspid and the parallelism of the dental axes will also be taken into account. Evaluations will be made by very precise radiological analysis using 3D CT-scan. Examinations will be done before and after closure of the extraction sites and will assess treatment efficacy using skeletal anchorage versus dental anchorage. Patients will also be requested to complete a satisfaction questionnaire. The study will comprise an inclusion appointment during which patient consent will be obtained and a regular monthly appointment during the 8 months of active treatment and space closure.

ELIGIBILITY:
Inclusion criteria:

* Aged from 12 to 50 years old
* Patient need orthodontic treatment with extraction of 2 maxillary bicuspid
* Patient has signed informed consent

Exclusion criteria:

* Patient younger than 12 and older than 50 years old
* Patient without social security affiliation
* Patient with a medical condition that indicates against orthodontic treatment

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

PRIMARY OUTCOMES:
We measure space extraction close after 8 months treatment. Angle class I cuspid and the parallelism of the dental axes will also be taken into account. | 8 months

SECONDARY OUTCOMES:
MINISCREW stability | 8 months
Anchorage teeth stability | 8 months
Success and Failure implantation percentage | 8 months
MINISCREW surgery difficulty | during the surgery act
Patient satisfaction | at 1 month and at 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Miller, Dentist, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; Claire Haignere, Dentist, Study Chair — Assistance Publique Hopitaux de Paris; Anne-Charlotte Six, Dentist, Study Chair — Assistance Publique Hopitaux de Paris; Alain Decker, Dentist, PhD, Study Chair — Assistance Publique Hopitaux de Paris
Locations (1):
- Bretonneau Hospital, Paris, France